CLINICAL TRIAL: NCT00615602
Title: A Multicenter Randomized Phase III Study Comparing 6 Versus 12 Months of Trastuzumab in Combination With Dose Dense Docetaxel Following FE75C as Adjuvant Treatment of Women With Axillary Lymph Node Positive Breast Cancer Over-expressing HER2
Brief Title: Six vs 12 Months of Trastuzumab With Docetaxel Following FEC as Adjuvant Treatment in N+ Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/04.23
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Axillary node positive; HER2 overexpression; Adjuvant chemotherapy; Dose dense; Docetaxel; Trastuzumab; FEC
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Trastuzumab; Epirubicin; Cyclophosphamide; Fluorouracil; Granulocyte Colony-Stimulating Factor; Lenograstim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): FEC -> TXT+H 12m
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: 5-fluoruracil; Drug: Granulocyte-colony stimulating growth factor
- 2 (Experimental): FEC -> TXT+H 6m
  Interventions: Drug: Docetaxel; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: 5-fluoruracil; Drug: Granulocyte-colony stimulating growth factor; Drug: Trastuzumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 as an IV infusion over 1h every two weeks for 4 cycles
  Other Names: Taxotere
Drug: Trastuzumab — Trastuzumab 6 mg/Kg IV over 30 min every two weeks for 4 cycles. Subsequently,trastuzumab 6 mg/Kg IV over 30 min for 12 months
  Other Names: Herceptin
  Arms: 1
Drug: Epirubicin — Epirubicin 75 mg/m2 IV push on day 1 every 2 weeks for 4 cycles
  Other Names: Farmorubicin
Drug: Cyclophosphamide — Cyclophosphamide 700 mg/m2 IV push on day 1 every 4 weeks
  Other Names: Endoxan
Drug: 5-fluoruracil — 5-fluoruracil 700 mg/m2 IV push on day 1 every 4 weeks
  Other Names: 5-FU
Drug: Granulocyte-colony stimulating growth factor — rhG-CSF 5 μg/kg/d on days 3-10 after each cycle
  Other Names: Granocyte; Neulasta
Drug: Trastuzumab — Trastuzumab 6mg/Kg IV over 30 min every 2 weeks for 4 cycles. Subsequently, trastuzumab 6mg/Kg IV over 30 min for 6 months
  Other Names: Herceptin
  Arms: 2

SUMMARY:
This trial will compare 6 versus 12 months of trastuzumab in combination with dose dense docetaxel following FE75C as adjuvant chemotherapy in women with axillary lymph node positive breast cancer overexpressing HER2

DETAILED DESCRIPTION:
Anthracycline-containing regimens are recommended as adjuvant treatment for women with node positive breast cancer. In at least three large randomized clinical trials the addition or sequential administration of a taxane (paclitaxel or docetaxel) to an antracycline-based regimen resulted in superior clinical outcome for women with node positive early breast cancer. In two large randomized studies the dose dense administration with G-CSF support of anthracycline-based and paclitaxel combination was superior to the same regimen administered every three weeks without growth factors as adjuvant therapy in women with axillary node positive breast cancer. In one randomized trial, docetaxel was proved superior to paclitaxel in women with metastatic breast cancer. Trastuzumab (anti-HER2 monoclonal antibody) in combination with paclitaxel was superior to paclitaxel alone in women with metastatic breast cancer overexpressing HER2

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically-confirmed unilateral invasive ductal or lobular breast adenocarcinoma
* HER2/c-neu over expression should be documented by either immunohistochemistry (score 3+) or FISH/CISH positivity. A score of 2+ by immunohistochemistry is acceptable only if FISH/CISH positive
* Within 60 days after the surgical excision of the primary tumor with tumor-free operation margins; at least 10 axillary lymph nodes have to be removed.
* Tumor involvement of at least one axillary lymph node (N0 with HER2/c-neu over expression are also eligible)
* Absence of any clinical or radiological evidence of local or metastatic disease
* Premenopausal or postmenopausal women aged 18-75 years old
* Adequate bone marrow function (absolute neutrophil count >1500/mm3, platelet count >100.000/mm3, hemoglobin >10gr/mm3)
* Adequate liver (bilirubin <1.0 times upper limit of normal and SGOT/SGPT <2.5 times upper limit of normal) and renal function (creatinine <1.5mg/dl)
* Adequate cardiac function (LVEF>50%). Normal electrocardiogram and absence of significant heart disease
* Written informed consent

Exclusion Criteria:

* Positive pregnancy test.
* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness.
* Prior or concurrent antineoplastic therapy e.g. hormonal therapy, radiation therapy, chemotherapy, biological agents.
* Previous history of other invasive malignancy other than non-melanomatous skin cancer.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2004-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Recurrence rate | Relapses by the time of 3-years follow up
Τoxicity profile | Toxicity assessment on each chemotherapy cycle
Quality of life between the two treatment arms | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki